CLINICAL TRIAL: NCT02496962
Title: Protective Effect of Statin on Arrhythmia and Heart Rate Variability in Healthy People With 48 Hours of Sleep Deprivation
Brief Title: Protective Effect of Statin on Sleep Deprivation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yang (Other)
Responsible Party: Sponsor-Investigator, Shi Yang, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2015-091-01
Record Dates: First submitted 2015-07-05; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin group (Experimental): drug: atorvastatin (Pfizer, U.S.); the frequency: 20mg atorvastatin was taken daily; duration: Study treatment was commenced 3 days before sleep deprivation and continued for 2 days during sleep deprivation.
  Interventions: Drug: Atorvastatin
- Control group (Placebo Comparator): drug: placebo (Pfizer, U.S.); the frequency: Placebo was taken daily; duration: Study treatment was commenced 3 days before sleep deprivation and continued for 2 days during sleep deprivation.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin were taken daily for 5 days
  Other Names: Lipitor
  Arms: Statin group
Drug: placebo — placebo were taken daily for 5 days
  Arms: Control group

SUMMARY:
This study aimed to investigate the effect of 48-h sleep deprivation on heart rate variability (HRV) in young healthy people and the protective effect of statin on arrhythmia and HRV.

DETAILED DESCRIPTION:
In the setting of earthquakes, floods, or fire disasters, rescue workers usually carry out their work without sleep. Sleep deprivation (SD), which is a strong stressor, can exert a large effect on the cardiovascular system of rescue workers. It has been reported that SD is associated with arrhythmia, dyslipidemia and type 2 diabetes. Heart rate variability (HRV) is acknowledged as a reliable marker of cardiac autonomic control, and the frequency of premature ventricular complexes can be an indicator of arrhythmogeneity. The investigators found that HRV was significantly decreased after 24-h sleep deprivation. Metoprolol could improve HRV and reduce the frequency of premature atrial and ventricular complexes. But sleepiness and hypotension occurred frequently in subjects treated with metoprolol. Statins have significant cardiovascular protective effects in patients with cardiovascular disease. Statin not only could regulate serum lipid level, but also have antioxidant and anti-inflammatory properties. This study aimed to investigate (1) the changes in heart rate variability and occurrence of cardiac arrhythmia by continuous ambulatory electrocardiogram (ECG) in young, healthy subjects undergoing 48h SD and (2) the effects of statin on HRV and arrhythmia after this agent was administered prophylactically before SD.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without cardiovascular disease

Exclusion Criteria:

* hypertension
* diabetes mellitus
* hyperthyroidism
* taking medication known to affect cardiovascular, metabolic, gastrointestinal, or immune function
* depression
* anxiety disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
a change in low-frequency (LF)/ high frequency (HF) | 48-h sleep deprivation
  The primary efficacy endpoint was the effect of statin on LF/HF measured by continuous ambulatory electrocardiogram monitoring after 48-h sleep deprivation.

SECONDARY OUTCOMES:
a change in the frequency of premature atrial and ventricular complexes | 48-h sleep deprivation
  The frequency of premature atrial and ventricular complexes during 48-h sleep deprivation were measured by continuous ambulatory electrocardiogram monitoring
a change in serum total cholesterol level | 48-h sleep deprivation
  serum total cholesterol level was measured after 48-h sleep deprivation
a change in serum high sensitivity C-reactive protein level | 48-h sleep deprivation
  serum high sensitivity C-reactive protein level was measured after 48-h sleep deprivation
a change in serum superoxide dismutase level | 48-h sleep deprivation
  serum superoxide dismutase level was measured after 48-h sleep deprivation

OTHER OUTCOMES:
a composite outcome (the incidences of treatment-emergent adverse events) | 48-h sleep deprivation
  Treatment-emergent adverse events (TEAEs): abnormal liver function, renal insufficiency and constipation

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Roost M, Nilsson P. [Sleep disorders--a public health problem. Potential risk factor in the development of type 2 diabetes, hypertension, dyslipidemia and premature aging]. Lakartidningen. 2002 Jan 17;99(3):154-7. Swedish. PMID 11838069
- [Background] Kumagai K. [Upstream therapy for atrial fibrillation]. Nihon Rinsho. 2013 Jan;71(1):86-90. Japanese. PMID 23631177
- [Background] Jacob KA, Nathoe HM, Dieleman JM, van Osch D, Kluin J, van Dijk D. Inflammation in new-onset atrial fibrillation after cardiac surgery: a systematic review. Eur J Clin Invest. 2014 Apr;44(4):402-28. doi: 10.1111/eci.12237. Epub 2014 Jan 30. PMID 24387767
- [Result] Chen WR, Shi XM, Yang TS, Zhao LC, Gao LG. Protective effect of metoprolol on arrhythmia and heart rate variability in healthy people with 24 hours of sleep deprivation. J Interv Card Electrophysiol. 2013 Apr;36(3):267-72; discussion 272. doi: 10.1007/s10840-012-9728-8. Epub 2012 Nov 20. PMID 23179915
- [Derived] Chen WR, Liu HB, Sha Y, Shi Y, Wang H, Yin DW, Chen YD, Shi XM. Effects of Statin on Arrhythmia and Heart Rate Variability in Healthy Persons With 48-Hour Sleep Deprivation. J Am Heart Assoc. 2016 Oct 31;5(11):e003833. doi: 10.1161/JAHA.116.003833. PMID 27799236